CLINICAL TRIAL: NCT01446796
Title: Hemodynamic and Clinical Effects of Continuous Right Ventricular Pacing in the Early Post-operative Period After Left Ventricular Assist Device Implantation
Brief Title: Right Ventricular (RV) Pacing in Early Post-operative Continuous Flow Left Ventricular Assist Device (LVAD)
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Recruitment futility
Sponsor: Duke University (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00026676
Record Dates: First submitted 2011-09-14; First posted 2011-10-05 (Estimated); Results first posted 2013-11-07 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure
Keywords: Ventricular assist device
MeSH Terms: conditions — Heart Failure | interventions — Defibrillators, Implantable

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Native Conduction (Placebo Comparator): Devices will be programmed to continuous atrial pacing at an AAI (atrial inhibited pacing) setting with base rate 90 bpm. Patients will not receive ventricular pacing.
  Interventions: Device: Implantable Cardioverter-Defibrillator (subject's pre-existing ICD)
- Continuous RV Pacing (Experimental): Devices will be programmed to continuous dual chamber pacing at a DDD (dual chamber dual pacing) setting with base rate ≥ 90 bpm (not to exceed 100 bpm) to achieve a majority (>80%) of paced right ventricular beats
  Interventions: Device: Implantable Cardioverter-Defibrillator (subject's pre-existing ICD)

INTERVENTIONS:
Device: Implantable Cardioverter-Defibrillator (subject's pre-existing ICD) — Pacing parameters set to AAI 90
  Arms: Native Conduction
Device: Implantable Cardioverter-Defibrillator (subject's pre-existing ICD) — Pacing parameters set to DDD 90-100
  Arms: Continuous RV Pacing

SUMMARY:
Continuous right ventricular (RV) pacing demonstrates harm in patients with normal left ventricular (LV) function as well as in patients with cardiomyopathy and clinical heart failure. However, little is known about RV pacing in patients with advanced heart failure treated with an implantable left ventricular assist device (LVAD). The univentricular support provided by contemporary continuous flow LVAD's has improved outcomes for many advanced heart failure patients, yet the incidence of RV failure in the early post-operative period following implantation is associated with significantly reduced survival and increased length of stay. Acute LVAD unloading of the left ventricle has adverse effects on RV shape and size that contribute to post-operative RV failure. By promoting RV synchrony, RV overdrive pacing may counteract these adverse mechanical alterations, improving RV systolic function and ultimately LVAD function.

The investigators will recruit all patients referred for an implantable, continuous flow LVAD at Duke University Medical Center who have an existing implantable dual-chamber cardioverter-defibrillator. Patients will be prospectively randomized into two cohorts to compare continuous right ventricular pacing vs. native ventricular conduction at equivalent heart rates. Multiple clinical outcomes will be examined over a two week period post-operatively including invasive hemodynamics, vasoactive medication use, end-organ function, RV function by Echocardiography as well as patient symptoms and functional status.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old, both men and women
* Existing implantable cardioverter-defibrillator (ICD)
* Referred for implantation of a continuous flow LVAD

Exclusion Criteria:

* Permanent left ventricular epicardial defibrillator in place
* Congenital heart disease with single ventricle physiology
* Right ventricular assist device (RVAD) in place
* Existing pacing indication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Rogers, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject provided initial consent but withdrew his consent prior to undergoing left ventricular assist device implantation. No further research activities for the study were performed with respect to this subject.
Period: Overall Study
Arm/Group | Continuous RV Pacing | Native Conduction
Started | 3 | 0
Completed | 2 (1. Study terminated early 2. One subject of three withdrew prior to randomization and did not start) | 0 (Study terminated early)
Not Completed | 1 | 0
Not completed — Withdrawal by Subject | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study terminated early
Groups:
- Continuous RV Pacing: Study terminated early due to recruitment
Arm/Group | Continuous RV Pacing
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 68 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Length of Hospitalization
Description: To determine whether continuous RV pacing reduces ICU length of stay (number of days) and overall hospital length of stay (number of days) post-LVAD implantation.
Time Frame: 14 days
Population: Study terminated early
Arm/Group | Native Conduction | Continuous RV Pacing
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Post-operative Need for Hemodynamic / Respiratory Support
Description: To determine whether continuous RV pacing reduces the need for inotropic / vasoactive agents, mechanical ventilation, or other circulatory support in the early post-operative period. Measured by the number of hemodynamic and respiratory support interventions and duration of those interventions.
Time Frame: 14 days
Population: Study terminated early due to low accrual. No data analysis completed.
Arm/Group | Continuous RV Pacing | Native Conduction
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Right Ventricular Function
Description: To determine whether continuous RV pacing improves invasive and non-invasive measures of RV function in the early period post-LVAD implantation. Measured by Pulmonary Artery catheter measures of intra-cardiac pressures and cardiac output in the ICU setting and by qualitative and quantitative Echocardiographic measures of RV function during the hospital course.
Time Frame: 14 days
Population: Study terminated early due to low accrual. No data analysis completed.
Arm/Group | Native Conduction | Continuous RV Pacing
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Functional Capacity and Symptoms
Description: To determine whether continuous RV pacing improves functional capacity and symptoms as measured by six minute walk test and symptoms questionnaires in the early post-LVAD implantation period.
Time Frame: 14 days
Population: Study terminated early due to low accrual. No data analysis completed.
Arm/Group | Native Conduction | Continuous RV Pacing
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Native Conduction | Continuous RV Pacing
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/2
Other Adverse Events (participants affected / at risk) | 0/0 | 0/2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes